CLINICAL TRIAL: NCT00720512
Title: AN OPEN-LABEL, MULTICENTER, RANDOMIZED PHASE III STUDY OF SECOND-LINE CHEMOTHERAPY WITH OR WITHOUT BEVACIZUMAB IN METASTATIC COLORECTAL CANCER PATIENTS WHO HAVE RECEIVED FIRST-LINE CHEMOTHERAPY PLUS BEVACIZUMAB.
Brief Title: Second-Line Combination Chemotherapy With or Without Bevacizumab in Treating Patients With Metastatic Colorectal Cancer Who Have Received First-Line Chemotherapy and Bevacizumab
Acronym: BEBYP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Gruppo Oncologico del Nord-Ovest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000598567; GONO-BEBYP-ASL607LIOM03; GONO-AIFA - FARM5C4FB4; EUDRACT:2007-002886-11
Record Dates: First submitted 2008-07-19; First posted 2008-07-22 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the colon; adenocarcinoma of the rectum; recurrent colon cancer; recurrent rectal cancer; stage IV colon cancer; stage IV rectal cancer; stage III rectal cancer; stage III colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Bevacizumab; Fluorouracil; Irinotecan; Leucovorin; Oxaliplatin

ARMS (2):
- Arm I (Active Comparator): Patients receive either irinotecan hydrochloride over 1 hour or oxaliplatin over 1 hour on day 1. Patients also receive leucovorin calcium IV over 2 hours and fluorouracil IV over 46 hours continuously beginning on day 1. Treatment repeats every 2 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: fluorouracil; Drug: irinotecan hydrochloride; Drug: leucovorin calcium; Drug: oxaliplatin
- Arm II (Experimental): Patients receive combination chemotherapy as in arm I and bevacizumab IV on day 1. Treatment repeats every 2 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab; Drug: fluorouracil; Drug: irinotecan hydrochloride; Drug: leucovorin calcium; Drug: oxaliplatin

INTERVENTIONS:
Biological: bevacizumab — Given IV
  Arms: Arm II
Drug: fluorouracil — Given IV
Drug: irinotecan hydrochloride — Given IV
Drug: leucovorin calcium — Given IV
Drug: oxaliplatin — Given IV

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irinotecan, oxaliplatin, leucovorin, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. It is not yet known whether combination chemotherapy is more effective with or without bevacizumab in treating metastatic colorectal cancer.

PURPOSE: This randomized phase III trial is studying second-line combination chemotherapy to see how well it works compared with or without bevacizumab in treating patients with metastatic colorectal cancer who have received first-line chemotherapy and bevacizumab.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the progression-free survival of second-line chemotherapy with or without bevacizumab in patients with metastatic colorectal cancer who have received first-line chemotherapy with bevacizumab.

Secondary

* To compare the overall survival, response rate, and safety profile of second-line chemotherapy of these regimens in these patients.
* To conduct pharmacogenomics assessment of candidate variants in the VEGF gene and evaluate their association with progression-free survival and other study outcomes.

OUTLINE: This is a multicenter study. Patients are stratified according to participating center, ECOG performance status (0 vs 1-2), disease-free interval from the last administration of first-line chemotherapy for metastatic disease (≤ 3 months vs > 3 months), and type of second-line chemotherapy (irinotecan hydrochloride, leucovorin calcium, and fluorouracil [FOLFIRI] vs oxaliplatin, leucovorin calcium, and fluorouracil [mFOLFOX-6]). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive either irinotecan hydrochloride over 1 hour or oxaliplatin over 1 hour on day 1. Patients also receive leucovorin calcium IV over 2 hours and fluorouracil IV over 46 hours continuously beginning on day 1.
* Arm II: Patients receive combination chemotherapy as in arm I and bevacizumab IV on day 1.

Treatment in both arms repeats every 2 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.

Existing formalin-fixed paraffin-embedded tumor tissue samples are assessed for pharmacogenomics and markers predictive of response, resistance to, or toxicity from bevacizumab. Samples are analyzed via RT-PCR, array comparative genomic hybridization, fluorescence in situ hybridization, sequencing of candidate genes, and immunohistochemistry.

After completion of study treatment, patients are followed for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colorectal adenocarcinoma

  * Metastatic or unresectable disease
* Progressive disease based on the following criteria:

  * Progression during or after first-line chemotherapy for metastatic disease, including any of the following:

    * Fluoropyrimidine-based monotherapy with bevacizumab
    * Fluoropyrimidine and irinotecan hydrochloride-based doublet with bevacizumab
    * Fluoropyrimidine and oxaliplatin-based doublet with bevacizumab
  * Progression after more than 3 months from the last administration of first-line chemotherapy for metastatic disease with a fluoropyrimidine, irinotecan hydrochloride, and oxaliplatin triplet (FOLFOXIRI) with bevacizumab to which the patient had previously responded
* Measurable disease, as assessed by RECIST criteria
* No prior or concurrent CNS metastasis

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 3 months
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL
* INR ≤ 1.5 times upper limit of normal (ULN)
* aPTT ≤ 1.5 ULN
* Serum bilirubin ≤ 1.5 times ULN
* AST and ALT ≤ 2.5 times ULN (< 5 times ULN if liver metastases present)
* Alkaline phosphatase ≤ 2.5 times ULN (< 5 times ULN if liver metastases present)
* Serum creatinine ≤ 1.5 times ULN
* Proteinuria < 2+ OR protein ≤ 1g by 24-hour urine
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No bowel obstruction or subobstruction
* No history of inflammatory enteropathy
* No prior extensive intestinal resection (i.e., > hemicolectomy or extensive small intestine resection with chronic diarrhea)
* No symptomatic peripheral neuropathy > grade 2
* No active uncontrolled infection
* No active disseminated intravascular coagulation
* No prior or concurrent malignancy, except for curatively treated basal cell and squamous cell carcinoma of the skin, or in situ carcinoma of the cervix
* No clinically significant cardiovascular disease, including any of the following:

  * Cerebrovascular accident within the past 6 months
  * Myocardial infarction within the past 6 months
  * Unstable angina
  * NYHA class II-IV chronic heart failure
  * Uncontrolled arrhythmia
* No uncontrolled hypertension
* No thromboembolic or hemorrhagic events within the past 6 months
* No evidence of bleeding diathesis or coagulopathy
* No serious, non healing wound/ulcer or serious bone fracture
* No significant traumatic injury within the past 28 days

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 6 weeks since prior radiotherapy
* At least 4 weeks since prior surgery
* No prior first-line chemotherapy for metastatic disease without bevacizumab
* No prior cetuximab or other investigational agents
* More than 28 days since prior open biopsy
* More than 28 days since prior and no concurrent major surgical procedure
* No concurrent therapeutic anticoagulation, antiplatelet agents, or NSAID with anti-platelet activity

  * Acetylsalicylic acid ≤ 325 mg/day allowed

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2008-06; Primary Completion 2013-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | last progression of the last patient

SECONDARY OUTCOMES:
Overall survival | the end of the stady
Response rate | last visit of the last patient
Safety | the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Falcone, MD, Principal Investigator — Presidio Ospedaliero di Livorno
Locations (21):
- Italy (21):
  - Universita Politecnica Delle Marche, Ancona
  - Azienda Usl 8 Arezzo, Arezzo
  - Ospedale degli Infermi - ASL 12, Biella
  - A. Perrino Hospital, Brindisi
  - Azienda Ospedaliera S. Elia, Caltanissetta
  - Ospedale Santa Croce, Cuneo
  - Ospedale San Giuseppe, Empoli
  - Ospedale E. Profili, Fabriano
  - Ospedale Civile S. Croce, Fano
  - Azienda Ospedaliera di Firenze, Florence
  - Azienda Ospedaliero Careggi, Florence
  - Istituto Nazionale per la Ricerca sul Cancro, Genoa
  - Ospendale S. Andrea EST, La Spezia
  - Azienda Ospedaliera Vito Fazzi, Lecce
  - Azienda USL12 Versilia, Lido di Camaiore
  - Ospedale Campo Di Marte Lucca, Lucca
  - Azienda Ospedaliera Maggiore Della Carita, Novara
  - Azienda Ospedaliera Pisana, Pisa
  - Arcispedale S. Maria Nuova, Reggio Emilia
  - Azienda Ospedaliera Universitaria Senese, Siena
  - Dipartimento Oncologico, Siena

REFERENCES:
- [Derived] Masi G, Salvatore L, Boni L, Loupakis F, Cremolini C, Fornaro L, Schirripa M, Cupini S, Barbara C, Safina V, Granetto C, Fea E, Antonuzzo L, Boni C, Allegrini G, Chiara S, Amoroso D, Bonetti A, Falcone A; BEBYP Study Investigators. Continuation or reintroduction of bevacizumab beyond progression to first-line therapy in metastatic colorectal cancer: final results of the randomized BEBYP trial. Ann Oncol. 2015 Apr;26(4):724-730. doi: 10.1093/annonc/mdv012. Epub 2015 Jan 18. PMID 25600568